CLINICAL TRIAL: NCT00542386
Title: A Phase III, Multi-centre, Double-blind, Randomised, Placebo-controlled Multiple Fixed-dose Study of MCI-196 Versus Placebo in Chronic Kidney Disease Stage V Subjects on Dialysis With Hyperphosphatemia and Dyslipidaemia (Incorporating Two Parallel High Dose Groups)
Brief Title: A Study of MCI-196 in Chronic Kidney Disease Subjects on Dialysis With Hyperphosphatemia and Dyslipidaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI-196-E08
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Dialysis; Hyperphosphatemia; Dyslipidemia
Keywords: Chronic Kidney Disease; Dialysis; Hyperphosphatemia; Dyslipidemia; Phosphate binder
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia; Dyslipidemias | interventions — cholebine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MCI-196
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCI-196 — 3g to 15g/day (3 times a day), Tablet, 12 weeks of fixed dose of study
  Other Names: Colestilan(INN),; Colestimide(JAN); CHOLEBINE®; BindRen®
  Arms: 1
Drug: Placebo — 3g to 15g/day (3 times a day), Tablet, 12 weeks of fixed dose of study
  Arms: 2

SUMMARY:
This is a phase III multi-centre study in two periods: the first period is a phosphate binder and lipid lowering drugs washout for 8 weeks, the second period is a double-blind, randomised, parallel group, fixed dose, for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or over
* Clinically stable haemodialysis or peritoneal dialysis
* Stable phosphate control
* On a stabilised phosphorus diet
* Female and of child-bearing potential have a negative serum pregnancy test
* Male subjects must agree to use appropriate contraception

Exclusion Criteria:

* Current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose them to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* A a serum albumin level<30.0g/L
* A PTH level >1000pg/mL
* A body mass index (BMI)<= 16.0kg/㎡ or =>40.0kg/㎡
* A serum LDL-C level >4.94mmol/L(190mg/dL)
* A serum triglycerides level >6.76mmol/L (600mg/dL)
* A History of significant gastrointestinal motility problems
* A positive test for HIV 1 and 2 antibodies
* A history of substance or alcohol abuse within the last year
* Seizure disorders
* A history of drug or other allergy
* A temporary catheter as a vascular access
* Participated in a clinical study with any experimental medication in the last 30 days or an experimental biological product within the last 90 days prior to signing of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2007-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma Europe
Locations (73):
- Hungary (7):
  - Ajka
  - Baja
  - Budapest
  - Esztergom
  - Győr
  - Hatvan
  - Kisvárda
- Italy (4):
  - Lecco
  - Modena
  - Pavia
  - Roma
- Malaysia (11):
  - Alor Star
  - Ipoh
  - Kajang
  - Klang
  - Kota Kinabalu
  - Kuala Terengganu
  - Kuantan
  - Kuching
  - Malacca
  - Seremban
  - Taiping
- Skopje, North Macedonia
- Poland (7):
  - Lodz
  - Poznan
  - Płock
  - Rybnik
  - Warsaw
  - Wroclaw
  - Zielona Góra
- Russia (29):
  - Arkhangelsk
  - Armavir
  - Chelyabinsk
  - Chita
  - Irkutsk
  - Ivanovo
  - Kaluga
  - Kemerovo
  - Khabarovsk
  - Krasnodar
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Novokuznetsk
  - Novorossiysk
  - Novosibirsk
  - Omsk
  - Petrozavodsk
  - Rostov-on-Don
  - Saint Petersburg
  - Smolensk
  - Tomsk
  - Tver'
  - Tyumen
  - Vladimir
  - Vladivostok
  - Volzhskiy
  - Yaroslavl
  - Yekaterinburg
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- Ukraine (10):
  - Chernivtsi
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Mykolaiv
  - Ternopil
  - Uzhhorod
  - Zaporizhya
  - Zhytomyr

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-196: 3 g: MCI-196: 3 g/ day
- MCI-196: 6 g: MCI-196: 6 g/ day
- MCI-196: 9 g: MCI-196: 9 g/ day
- MCI-196: 12 g: MCI-196: 12 g/ day
- MCI-196: 15 g: MCI-196: 15 g/ day
- Pooled Placebo: Placebo 9 tablets, 12 tablets and 15 tablets/ day
Period: Overall Study
Arm/Group | MCI-196: 3 g | MCI-196: 6 g | MCI-196: 9 g | MCI-196: 12 g | MCI-196: 15 g | Pooled Placebo
Started | 104 | 102 | 99 | 103 | 102 | 132
Completed | 61 | 74 | 66 | 65 | 62 | 82
Not Completed | 43 | 28 | 33 | 38 | 40 | 50
Not completed — Adverse Event | 1 | 7 | 7 | 8 | 13 | 4
Not completed — Death | 0 | 0 | 1 | 2 | 1 | 2
Not completed — Lack of Efficacy | 32 | 12 | 10 | 13 | 7 | 31
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 5 | 8 | 10 | 11 | 15 | 7
Not completed — Other Reasons | 4 | 1 | 4 | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Each one subject in the MCI-196 9 g group, MCI-196 12 g group, and MCI-196 15 g group were randomised but did not receive any study medication. Therefore these 3 subjects were excluded in the baseline characteristics analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-196: 3 g | MCI-196: 6 g | MCI-196: 9 g | MCI-196: 12 g | MCI-196: 15 g | Pooled Placebo | Total
Number analyzed (Participants) | 104 | 102 | 98 | 102 | 101 | 132 | 639
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (12.20) | 48.7 (14.64) | 47.3 (12.55) | 49.5 (12.41) | 50.7 (11.34) | 48.5 (12.54) | 49.1 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 54 | 48 | 48 | 46 | 55 | 299
  Male | 56 | 48 | 50 | 54 | 55 | 77 | 340

OUTCOME MEASURES:

1. Primary Outcome: The Change in Serum Phosphorus
Description: The change from baseline to week 12
Time Frame: 12 weeks
Population: ITT: The ITT population included all subjects who received a randomisation number, took study medication, and had at least 1 central laboratory serum phosphorus or LDL-C value after the start
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MCI-196: 3 g | MCI-196: 6 g | MCI-196: 9 g | MCI-196: 12 g | MCI-196: 15 g | Pooled Placebo
Number analyzed (Participants) | 104 | 101 | 97 | 100 | 99 | 130
mg/dL | -0.23 (1.62) | -0.77 (1.97) | -0.97 (1.68) | -0.71 (1.84) | -1.41 (1.43) | -0.12 (1.70)

2. Primary Outcome: The Change in LDL-cholesterol
Description: The percentage change from baseline to week 12
Time Frame: 12 weeks
Population: ITT: The ITT population included all subjects who received a randomisation number, took study medication, and had at least 1 central laboratory serum phosphorus or LDL-C value after the start of study medication.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MCI-196: 3 g | MCI-196: 6 g | MCI-196: 9 g | MCI-196: 12 g | MCI-196: 15 g | Pooled Placebo
Number analyzed (Participants) | 104 | 101 | 97 | 100 | 99 | 130
Percent change | -16.66 (20.05) | -23.56 (20.99) | -27.64 (21.45) | -29.44 (25.28) | -27.46 (24.57) | 2.77 (17.44)

3. Secondary Outcome: The Change in Total-cholesterol
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: The Change in HDL-cholesterol
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: The Change in Triglycerides
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: The Change in PTH
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: The Change in Ca
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: The Change in Ca x P Ion Product
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: The Incidence of Adverse Events
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Each one subject in the MCI-196 9 g group, MCI-196 12 g group, and MCI-196 15 g group were randomised but did not receive any study medication. Therefore these 3 subjects were excluded for the safety evaluation.
Arm/Group | MCI-196: 3 g | MCI-196: 6 g | MCI-196: 9 g | MCI-196: 12 g | MCI-196: 15 g | Pooled Placebo
Serious Adverse Events (participants affected / at risk) | 3/104 | 1/102 | 2/98 | 7/102 | 5/101 | 8/132
Other Adverse Events (participants affected / at risk) | 47/104 | 44/102 | 49/98 | 53/102 | 59/101 | 65/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196: 3 g (N=104) | MCI-196: 6 g (N=102) | MCI-196: 9 g (N=98) | MCI-196: 12 g (N=102) | MCI-196: 15 g (N=101) | Pooled Placebo (N=132)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site phlebitis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal transplant (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196: 3 g (N=104) | MCI-196: 6 g (N=102) | MCI-196: 9 g (N=98) | MCI-196: 12 g (N=102) | MCI-196: 15 g (N=101) | Pooled Placebo (N=132)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 2 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 6 | 6 | 2 | 5 | 4
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 4 | 0 | 4
Hypertonia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uraemic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Convulsions local (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tonic convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Injection site abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Vaginitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 2
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 4 | 1 | 3 | 3 | 4 | 1
Pyrexia (General disorders) | 4 | 1 | 1 | 0 | 1 | 1
Chills (General disorders) | 2 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 2 | 0 | 0 | 1
Malaise (General disorders) | 0 | 2 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catheter related complication (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Aortic valve calcification (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 6 | 4 | 5 | 7
Nausea (Gastrointestinal disorders) | 4 | 9 | 12 | 19 | 20 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 4 | 1 | 3 | 1
Frequent bowel movements (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 0 | 3 | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 8 | 7 | 5 | 9 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 6 | 0 | 5 | 2
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 8 | 11 | 6 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 2 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 2 | 7 | 6 | 4
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 0
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1 | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood parathyroid hormone increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 3
Blood pressure increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 1 | 0 | 2 | 1
Blood phosphorus increased (Investigations) | 3 | 0 | 1 | 1 | 0 | 3
Cardiac murmur (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Carotid bruit (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 1 | 2 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 1
Extensive interdialytic weight gain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 6 | 4 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 6 | 2 | 3
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 3 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased activity (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal transplant (Surgical and medical procedures) | 1 | 1 | 1 | 1 | 0 | 0
Nephrectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 1
Parathyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other